CLINICAL TRIAL: NCT02226692
Title: Risk of Poor Prognosis in Patients With Chronic Low Back Pain : Can it be Predicted by Physical Tests and Screening Tools ? - An Observational Study
Brief Title: Prognostic Factors of Disabling Low Back Pain in Patients With Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Université du Québec à Trois-Rivières (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Institut de Recherche Robert-Sauvé en Santé et en Sécurité du Travail (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Dr Martin Descarreaux DC, PhD, Université du Québec à Trois-Rivières
Other Study IDs: UQTR-2011-PFAC
Record Dates: First submitted 2014-08-12; First posted 2014-08-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Low Back Pain; Mechanical Low Back Pain
Keywords: chronic low back pain; prognostic factors; disabling low back pain; lumbar muscle activity; start back screening tool; physical evaluation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- nonspecific chronic low back pain: Physical examination and follow-up assessment by questionnaires at 2, 4, 6, and 12 months

SUMMARY:
The aim of the present study is to quantify the relative contribution of variables obtained during a physical fitness evaluation and a short screening questionnaire in determining the short-term and long term risk of persistent disabling low back pain in patients with chronic low back pain. It has been hypothesized that patients with higher physical fitness will present a lower risk of persistent disabling low back pain and so, a lower score on the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* adults between 18 and 60 years old
* nonspecific low back pain : pain located between the twelfth rib and the inferior gluteal fold for which no specific source of pain could be identified
* chronic low back pain : pain present for 12 weeks or more, and included both constant and recurrent patterns of pain
* able to read and understand French

Exclusion Criteria:

* History of surgery or major trauma to the spine
* Current use of medication known to impair physical effort and pain perception
* Lumbar scoliosis of more than 20°
* Collagenosis, severe osteoporosis
* Neuromuscular disease
* Malignant tumor
* Non-controlled hypertension
* Infection
* Radiculopathy
* Progressive neurologic defect
* Myelopathy
* Lumbar disc hernia
* Pregnancy
* Active lower body injury and/or severe and disabling pain limiting the capacity to undergo the evaluation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: volunteer with chronic nonspecific low back pain will be recruited among the university's community, its outpatients' chiropractic clinic and through advertisements in the local newspaper. They will first be screened by clinicians at the outpatients' chiropractic clinic in order to assess for the various inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Disability level | 2 months
  Oswestry disability index
Disability level | 4 months
  Oswestry disability index
Disability level | 6 months
  Oswestry disability index
Disability level | 12 months
  Oswestry disability index

SECONDARY OUTCOMES:
Pain intensity in the past 2 months | 2 months
  101 points numerical rating scale
Fear of movement level | 2 months
  Tampa scale for kinesiophobia
Patient's global impression of change from baseline | 6 months
  Patient's global impression of change scale
Patient's global impression of change from 6 months | 12 months
  Patient's global impression of change scale
Pain intensity in the past 2 months | 4 months
  101 points numerical rating scale
Pain intensity in the past 2 months | 6 months
  101 points numerical rating scale
Pain intensity in the past 6 months | 12 months
  101 points numerical rating scale
Pain intensity in the past week | 12 months
  101 points numerical rating scale
Fear of movement level | 4 months
  Tampa scale for kinesiophobia
Fear of movement level | 6 months
  Tampa scale for kinesiophobia
Fear of movement level | 12 months
  Tampa scale for kinesiophobia

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Université du Québec à Trois-Rivières, Trois-Rivières, Quebec, Canada

REFERENCES:
- [Derived] Page I, Abboud J, O Shaughnessy J, Laurencelle L, Descarreaux M. Chronic low back pain clinical outcomes present higher associations with the STarT Back Screening Tool than with physiologic measures: a 12-month cohort study. BMC Musculoskelet Disord. 2015 Aug 19;16:201. doi: 10.1186/s12891-015-0669-0. PMID 26286385